CLINICAL TRIAL: NCT02582333
Title: Clinical Course Study in Chronic Hepatitis B After Nucleos(t)Ide Analogue Therapy
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Teng-Yu Lee, Gastroenterology & Hepatology Division, Taichung Veterans General Hospital
Other Study IDs: CF15240B
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Virological Breakthrough; Prognosis
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HBV DNA and genotype
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tenofovir: Chronic hepatitis B patients who receive tenofovir as their first anti-HBV therapy and are indicated for stopping tenofovir therapy
  Interventions: Other: Observation for clinical and virological changes
- Entecavir: Chronic hepatitis B patients who receive entecavir as their first anti-HBV therapy and are indicated for stopping entecavir therapy
  Interventions: Other: Observation for clinical and virological changes

INTERVENTIONS:
Other: Observation for clinical and virological changes — Only observation after stopping nucleos(t)ide analogue

SUMMARY:
Background:

Taiwan is one of the area with the highest prevalence of chronic hepatitis B (CHB), and many patients die of hepatitis B virus (HBV)-related cirrhosis or liver cancer that have been the leading causes of death in Taiwan for many years. For effectively treating CHB, antiviral therapy for CHB has been reimbursed by the National Health Insurance in Taiwan since 1998, and nucleos(t)ide analogues (NAs) can be used for patients with active hepatitis B and high viral load in a maximum duration of three years. However, there is a significant proportion of patients suffering from hepatitis B recurrence after discontinuation of NA therapy, and hepatitis B recurrence may result in liver cirrhosis and liver cancer. To the best of current knowledge, in what conditions that the NA therapy can be successfully discontinued without hepatitis recurrence remain largely unclear. Therefore, this study is designed to evaluate the clinical and virological changes of CHB patients after stopping NA therapy, and finding the prognostic indicators may be an important basis for stopping NA therapy in CHB patients in the future.

Objectives:

1. To access the clinical and virological changes after stopping NA therapy
2. To determine important prognostic indicators for stopping NA therapy

Methods:

In this prospective cohort study, the investigators plan to recruit CHB patients who are indicated for stopping NA therapy in the outpatient clinics according to the inclusion and exclusion criteria of this study, and clinical and virological data will be collected during routine clinic visits after stopping NA therapy. Prognostic factors will be analyzed according the following data:

1. Patient characteristics: including age, sex, height, weight, waist circumference, history of alcohol drinking, antiviral therapy history, hepatitis history, and drug history.
2. Blood tests: During routine clinic visits and blood tests every 12 weeks or at hepatitis flare in the first 2 years after stopping NA therapy, liver function and virological status tests will be conducted for analysis.

DETAILED DESCRIPTION:
Background:

Taiwan is one of the area with the highest prevalence of chronic hepatitis B (CHB), and many patients die of hepatitis B virus (HBV)-related cirrhosis or liver cancer that have been the leading causes of death in Taiwan for many years. For effectively treating CHB, antiviral therapy for CHB has been reimbursed by the National Health Insurance in Taiwan since 1998, and nucleos(t)ide analogues (NAs) can be used for patients with active hepatitis B and high viral load in a maximum duration of three years. However, there is a significant proportion of patients suffering from hepatitis B recurrence after discontinuation of NA therapy, and hepatitis B recurrence may result in liver cirrhosis and liver cancer. To the best of current knowledge, in what conditions that the NA therapy can be successfully discontinued without hepatitis recurrence remain largely unclear. Therefore, this study is designed to evaluate the clinical and virological changes of CHB patients after stopping NA therapy, and finding the prognostic indicators may be an important basis for stopping NA therapy in CHB patients in the future.

Objectives:

1. To access the clinical and virological changes after stopping NA therapy
2. To determine important prognostic indicators for stopping NA therapy

Methods:

In this prospective cohort study, the investigators plan to recruit CHB patients who are indicated for stopping NA therapy in the outpatient clinics according to the inclusion and exclusion criteria of this study, and clinical and virological data will be collected during routine clinic visits after stopping NA therapy. Prognostic factors will be analyzed according the following data:

1. Patient characteristics: including age, sex, height, weight, waist circumference, history of alcohol drinking, antiviral therapy history, hepatitis history, and drug history.
2. Blood tests: During routine clinic visits and blood tests every 12 weeks or at hepatitis flare in the first 2 years after stopping NA therapy, liver function and virological status tests will be conducted for analysis.

Importance:

To clinicians in treating chronic hepatitis B, this study will provide important data regarding the clinical courses after stopping NA therapy, and important prognostic indicators may be determined. These findings could help clinicians in decision making for discontinuation of NA therapy and booking follow-up schedules. To basic scientists, this study will provide the virological changes after stopping NA therapy, and these findings may help developing further virological researches.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 20 years old
2. Chronic hepatitis B patients who received tenofovir or entecavir as their first anti-HBV therapy
3. Patients who have received nucleos(t)ide analogue therapy for > 3 years or reached the stopping criteria of APASL ( HBeAg+ patients: HBeAg seroconversion > 12 months; HBeAg - patients: HBV DNA undetectable > 12 months)

Exclusion Criteria:

1. History of liver cirrhosis or hepatocellular carcinoma
2. Recipients of liver transplantation
3. Concurrent malignancies (except curable skin cancers)
4. Concomitant use of immunosuppressants
5. Coinfection with HCV, HDV, HIV

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients who are indicated for stopping nucleos(t)ide analogue therapy in the outpatient clinics according to the inclusion and exclusion criteria of this study
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
HBsAg seroconversion | 2 years after stopping nucleos(t)ide analogue
  HBsAg negative, anti-HBs positive

CONTACTS AND LOCATIONS:
Overall Officials: Teng-Yu Lee, MD, PhD, Study Chair — Taichung Veterans General Hospital
Locations (4):
- Taiwan (4):
  - Show Chwan Memorial Hospital, Changhua
  - Cheng Ching General Hospital-Chung Kang Branch, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung